CLINICAL TRIAL: NCT03123978
Title: A Safety Trial of Enzalutamide in Combination With PDMX1001/Niclosamide in Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Enzalutamide and Niclosamide in Treating Patients With Recurrent or Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mamta Parikh (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pandomedx (Other)
Responsible Party: Sponsor-Investigator, Mamta Parikh, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 914328; UCDCC#264 (Other: UC Davis IRB); P30CA093373 (NIH); NCI-2017-00294 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
Keywords: castration resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (niclosamide, enzalutamide) (Experimental): Patients receive niclosamide PO BID and enzalutamide PO QD on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Drug: Niclosamide

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Drug: Niclosamide — Given PO

SUMMARY:
This phase I trial studies the best dose and side effects of niclosamide when given together with enzalutamide in treating patients with castration-resistant prostate cancer that has come back or has spread to other places in the body. Androgens can cause the growth of prostate cancer cells. Hormone therapy using enzalutamide may fight prostate cancer by lowering the amount of androgen the body makes and/or blocking the use of androgen by the tumor cells. Niclosamide may block signals that enhance prostate cancer cell growth. Giving enzalutamide and niclosamide may work better in treating patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of niclosamide (PDMX1001/niclosamide) and enzalutamide in patients with castration-resistant prostate cancer (CRPC).

II. To determine the recommended phase II dose (RP2D) of PDMX1001/niclosamide and enzalutamide for the treatment of patients with CRPC.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of PDMX1001/niclosamide. II. To determine the number of patients who have a prostate-specific antigen (PSA) response that is a 50% or more reduction from the baseline.

III. To identify overall responses as determined by the Prostate Cancer Working Group 2 (PCWG2) criteria.

IV. To evaluate the progression-free survival (PFS) of CRPC patients treated with PDMX1001/niclosamide and enzalutamide.

V. To evaluate molecular correlatives for patient response and outcomes through the analysis of patient baseline tumor specimens (diagnostic biopsy) along with serial blood specimens.

OUTLINE: This is a dose-escalation study of niclosamide.

Patients receive niclosamide orally (PO) twice daily (BID) and enzalutamide PO once daily (QD) on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed carcinoma of the prostate (CaP); CaP can be recurrent disease after definitive therapy (radical prostatectomy or radiation therapy) for localized CaP, or metastatic CaP
* Patients must have CaP deemed to be castration-resistant by one or more of the following criteria (despite androgen deprivation when applicable):

  * Progression of unidimensionally measurable disease assessed within 42 days prior to initial administration of drug
  * Progression of evaluable but not measurable disease assessed within 42 days prior to initial administration of drug for PSA evaluation and for imaging studies (e.g, bone scans)
  * Rising PSA, defined as at least two consecutive rises in PSA to be documented over a reference value (measure 1); the first rising PSA (measure 2) should be taken at least 7 days after the reference value; a third confirmatory PSA measure (2nd beyond the reference level) should be greater than the second measure, and it must be obtained at least 7 days after the 2nd measure; if this is not the case, a fourth PSA measurement is required to be taken and be greater than the second measure
* Measurable disease is not required:

  * Patients who have measurable disease must have had X-rays, computed tomography (CT) scans or physical examinations used for tumor measurement completed within 28 days prior to initial administration of drug
  * Patients must have non-measurable disease (such as nuclear medicine bone scans) and non-target lesions (such as PSA level) assessed within 28 days prior to initial administration of drug
  * Soft tissue disease that has been radiated within two months prior to registration is not assessable as measurable disease; soft tissue disease that has been radiated two or more months prior to registration is assessable as measurable disease provided that the lesion has progressed following radiation; as the biology of previously irradiated tumors may be different from non-irradiated tumors, patients must have at least one measurable lesion outside the previously irradiated region in order to be considered to have measurable disease
  * If PSA is the only indicator of disease without any evidence of metastasis, PSA value must be 5.0 or higher
* Expression of AR-V7 is not required as expression of AR-V7 can occur during enzalutamide and contribute to resistance to enzalutamide
* Patients must have been surgically or medically castrated; if the method of castration was luteinizing hormone-releasing hormone (LHRH) agonists (leuprolide or goserelin) or antagonists (degarelix), then the patient must be willing to continue the use of LHRH agonists or antagonists; serum testosterone must be at castration levels (< 50 ng/dL) within 3 months prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy should be deemed greater than 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of enzalutamide and PDMX1001/niclosamide administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have received any other investigational agents within the preceding 4 weeks
* Patients taking herbal or other alternative medicines for the treatment of prostate cancer, including but not limited to saw palmetto, prostate cancer (PC)-SPES
* Patient has received enzalutamide for the treatment of prostate cancer; however, previous treatment with other hormonal therapy (bicalutamide, flutamide, nilutamide, abiraterone and ketoconazole) or chemotherapy (docetaxel, cabazitaxel or mitoxantrone) is allowed
* Other malignancies within the past 3 years except for adequately treated basal or squamous cell carcinomas of the skin or other stage 0 or I cancers
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or PDMX1001/niclosamide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Patients with symptomatic metastatic prostate cancer experiencing moderate to severe pain, impaired organ function or spinal cord compression will be excluded from this study unless these issues have been addressed

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of grade 3 or higher assessed by National Cancer Institute Common Terminology Criteria for Adverse Events 4.0 | Up to 4 weeks
  Adverse events and adverse events of grade 3 or higher will be listed for each patient and summarized by body system in a frequency table.
RP2D of niclosamide and enzalutamide | Up to 2 years
  Determination of dose limiting toxicity as graded according to NCI CTCAE 4.0.

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  Will be estimated using the product-limit method of Kaplan and Meier; medians and 95% confidence intervals will be computed.
PFS | Up to 5 years
  Will be estimated using the product-limit method of Kaplan and Meier; medians and 95% confidence intervals will be computed.
Rate of PSA response which is defined as >= 50% decrease | Baseline up to 2 years
  The characteristics of the study participants will be summarized using frequencies and percentages for categorical variables and descriptive statistics (mean, standard deviation, median, minimum, maximum) for numeric variables. The proportion of participants who experience a PSA response will be computed, along with the exact 95% confidence interval.
Time to treatment failure | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier; medians and 95% confidence intervals will be computed.

OTHER OUTCOMES:
Analysis of laboratory correlatives | Up to 2 years
  Will be performed between patients who respond and those who do not respond, and between specimens obtained during response and those specimens obtained during resistance in the same patients. Will be descriptive and exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States